CLINICAL TRIAL: NCT00370292
Title: Pemetrexed Monochemotherapy in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer. A Pilot Study to Define the Best Dosing Schedule for a Planned Phase II Randomized Trial
Brief Title: Dosage Schedule Study of Pemetrexed Monochemotherapy for Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10940; H3E-IT-S105
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Results first posted 2009-10-12 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed - Before Protocol Amendment (Experimental)
  Interventions: Drug: Pemetrexed - Before Protocol Amendment
- Pemetrexed - After Protocol Amendment (Experimental)
  Interventions: Drug: Pemetrexed - After Protocol Amendment

INTERVENTIONS:
Drug: Pemetrexed - Before Protocol Amendment — 500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles or disease progression, unacceptable toxicity or patient decision to discontinue
  Other Names: LY231514; Alimta
  Arms: Pemetrexed - Before Protocol Amendment
Drug: Pemetrexed - After Protocol Amendment — 500 milligrams per square meter (mg/m2), intravenous (IV), every 21 days x 6 cycles or disease progression, unacceptable toxicity or patient decision to discontinue.
  Other Names: LY231514; Alimta
  Arms: Pemetrexed - After Protocol Amendment

SUMMARY:
Patients affected by non-small cell lung cancer (NSCLC) will be treated in pemetrexed monochemotherapy regimen for a maximum of 8 cycles. Pemetrexed is an enhancer of some biomolecules involved in the gemcitabine mechanism of action. Purpose of the trial is to monitor the blood values of these biomolecules at different time intervals, to optimize the synergism between pemetrexed and gemcitabine.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically proven IIIB and IV NSCLC.
* No symptomatic uncontrolled brain metastasis
* Not suitable for platinum containing regimens if chemo-naive
* Performance status less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Creatinine Clearance (CrCl) greater than or equal to 45 milliliters per min (mL/min)

Exclusion Criteria

* Prior radiation to greater than 25% of bone marrow
* Inability to interrupt Aspirin at doses of greater than 1.3 grams/day or non-steroidal anti-inflammatory agents for a 5-day period.
* Presence of clinically relevant third-space fluid collections not controllable.
* Significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan, Italy

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 19 enrolled patients, 12 were enrolled before the protocol amendment was made effective (i.e. 2-weekly administration) and 7 were enrolled after the amendment (i.e. 3-weekly administration).
Groups:
- Pemetrexed: 500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles (pre-amendement) or 21 days x 6 cycles (post-amendment) or disease progression, unacceptable toxicity or patient decision to discontinue.
Period: Overall Study
Arm/Group | Pemetrexed
Started | 19
Completed | 6
Not Completed | 13
Not completed — Disease Progression | 4
Not completed — Adverse Event | 7
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed - Before Amendment: 500 milligrams per square meter (mg/m2), intravenous (IV), every 14 days x 8 cycles or disease progression, unacceptable toxicity or patient decision to discontinue.
- Pemetrexed - After Amendment: 500 milligrams per square meter (mg/m2), intravenous (IV), every 21 days x 6 cycles or disease progression, unacceptable toxicity or patient decision to discontinue.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed - Before Amendment | Pemetrexed - After Amendment | Total
Number analyzed (Participants) | 12 | 7 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (10.34) | 69.4 (6.45) | 69.2 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 2 | 11
Region of Enrollment [Number; unit: participants]
  Italy | 12 | 7 | 19
Disease Stages [Number; unit: participants] — Stage means how big the tumor is and how far it's spread. Stages range from 0 (tumor has not spread) to IV (tumor has spread to other organs).
  participants
    Not Known | 0 | 1 | 1
    Stage IA | 2 | 0 | 2
    Stage IB | 1 | 0 | 1
    Stage IIA | 1 | 0 | 1
    Stage IIB | 0 | 1 | 1
    Stage IIIA | 0 | 1 | 1
    Stage IIIB | 3 | 2 | 5
    Stage IV | 5 | 2 | 7
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 4 | 1 | 5
    1 - Ambulatory, Restricted Strenuous Activity | 6 | 5 | 11
    2 - Ambulatory, No Work Activities | 2 | 1 | 3
Histopathological Grade [Number; unit: participants] — Assesses the extent to which cancer cells are similar in appearance and function to healthy cells of the same tissue type. Grades range from 1 (least aggressive and best prognosis) to 4 (most aggressive and worst prognosis).
  participants
    Not Done | 7 | 2 | 9
    G1 - Well-Differentiated | 1 | 1 | 2
    G2 - Moderately Differentiated | 2 | 1 | 3
    G3 - Poorly Differentiated | 2 | 3 | 5
Previous Anti-Tumor Treatment [Number; unit: participants]
  No | 5 | 1 | 6
  Yes | 7 | 6 | 13
Previous Surgery [Number; unit: participants] — Participants having surgery could have more than one type of surgery.
  participants
    Surgery - No | 4 | 1 | 5
    Surgery - Yes: Pneumonectomy | 0 | 1 | 1
    Surgery - Yes: Lobectomy | 3 | 3 | 6
    Surgery - Yes: Other | 5 | 3 | 8
    Surgery - Yes: Radical | 5 | 4 | 9
Race/Ethnicity [Number; unit: participants]
  Caucasian | 12 | 7 | 19
Tumor Type [Number; unit: participants]
  Adenocarcinoma | 5 | 6 | 11
  Squamous Cell Carcinoma | 5 | 1 | 6
  Other | 2 | 0 | 2
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic Blood Pressure (SBP) | 138.0 (13.17) | 146.9 (21.54) | 141.6 (17.08)
  Diastolic Blood Pressure (DBP) | 81.8 (7.97) | 83.6 (9.45) | 82.5 (8.37)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meters (m^2)] — BSA = 0.007184 x weight(kg)^0.425 x height(cm)^0.725
  square meters (m^2) | 1.7 (0.17) | 1.7 (0.13) | 1.7 (0.16)
Body Temperature [Mean (Standard Deviation); unit: degrees Celsius (°C)] | 36.1 (0.58) | 35.9 (0.36) | 36.0 (0.49)
Heart Rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 82.9 (14.98) | 78.6 (8.52) | 81.1 (12.58)
Height [Mean (Standard Deviation); unit: centimeters (cm)] — One participant in the Pemetrexed - Before Amendment group was missing a baseline height measurement.
  centimeters (cm) | 169.2 (10.15) | 162.1 (9.04) | 166.4 (10.09)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — One participant in the Pemetrexed - Before Amendment group was missing a baseline weight measurement.
  kilograms (kg) | 70.2 (15.28) | 66.3 (9.43) | 68.7 (13.13)

OUTCOME MEASURES:

1. Primary Outcome: Mean Deoxycytidine Kinase (dCK) Expression Evaluated at Cycle 1, Cycle 2, and Cycle 3
Description: dCK and hENT expression (see Outcome #2) on normal lymphocytes were measured after Pemetrexed administration to evaluate if there was reproducible timing of maximum dCK expression, and to assess proper time interval between pemetrexed and gemcitabine for treatment of patients with advanced Non-Small Cell Lung Cancer (NSCLC). Values are calculated as ratio between thereshold cycles (number of polymerase chain reaction [PCR] cycles) with respect to a reference gene; in this case glyceraldehyde 3-phosphate dehydrogenase (GAPDH).
Time Frame: pre-dose, 1, 2, 4, 6, 24, and 48 hours post-dose (3 cycles)
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mRNA relative values (ratio with GAPDH)
Groups:
- dCK - Cycle 1: Mean dCK expression evaluated at Cycle 1.
- dCK - Cycle 2: Mean dCK expression evaluated at Cycle 2.
- dCK - Cycle 3: Mean dCK expression evaluated at Cycle 3.
Arm/Group | dCK - Cycle 1 | dCK - Cycle 2 | dCK - Cycle 3
Number analyzed (Participants) | 19 | 19 | 19
mRNA relative values (ratio with GAPDH)
  Pre-Dose | 0.92 (0.03) | 0.92 (0.03) | 0.92 (0.02)
  1 Hour Post-Dose | 0.96 (0.04) | 0.95 (0.03) | 0.96 (0.03)
  2 Hours Post-Dose | 0.96 (0.04) | 0.96 (0.04) | 0.97 (0.02)
  4 Hours Post-Dose | 0.93 (0.04) | 0.94 (0.04) | 0.92 (0.03)
  6 Hours Post-Dose | 0.92 (0.03) | 0.91 (0.04) | 0.91 (0.03)
  24 Hours Post-Dose | 0.96 (0.04) | 0.97 (0.03) | 0.96 (0.03)
  48 Hours Post-Dose | 0.97 (0.04) | 0.96 (0.04) | 0.97 (0.03)
Statistical Analysis 1: Comparison: dCK - Cycle 1 vs dCK - Cycle 2 vs dCK - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 1 Hour Post-Dose (1 hour across cycles compared with pre-dose across cycles)
Statistical Analysis 2: Comparison: dCK - Cycle 1 vs dCK - Cycle 2 vs dCK - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 2 Hours Post-Dose (2 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 3: Comparison: dCK - Cycle 1 vs dCK - Cycle 2 vs dCK - Cycle 3; Test type: Superiority or Other; p = 0.030, Repeated Measures Analysis of Variance — P-value for 4 Hours Post-Dose (4 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 4: Comparison: dCK - Cycle 1 vs dCK - Cycle 2 vs dCK - Cycle 3; Test type: Superiority or Other; p = 0.166, Repeated Measures Analysis of Variance — P-value for 6 Hours Post-Dose (6 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 5: Comparison: dCK - Cycle 1 vs dCK - Cycle 2 vs dCK - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 24 Hours Post-Dose (24 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 6: Comparison: dCK - Cycle 1 vs dCK - Cycle 2 vs dCK - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 48 Hours Post-Dose (48 hours across cycles compared with pre-dose across cycles)

2. Secondary Outcome: Best Objective Tumor Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to measured response (every 14 days for 6 cycles)
Population: Number of participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed - Before Amendment | Pemetrexed - After Amendment
Number analyzed (Participants) | 12 | 7
participants
  Partial Response | 1 | 0
  Stable Disease | 2 | 4
  Progressive Disease | 3 | 0
  Early Death | 1 | 0
  Unconfirmed Stable Disease | 5 | 3

3. Primary Outcome: Mean Human Equilibrative Nucleoside Transporter 1 (hENT) Expression Evaluated at Cycle 1, Cycle 2, and Cycle 3
Description: dCK (see Outcome #1)and hENT expression (see Outcome #2) on normal lymphocytes were measured after Pemetrexed administration to evaluate if there was reproducible timing of maximum dCK expression, and to assess proper time interval between pemetrexed and gemcitabine for treatment of patients with advanced Non-Small Cell Lung Cancer (NSCLC). Values are calculated as ratio between thereshold cycles (number of polymerase chain reaction [PCR] cycles) with respect to a reference gene; in this case glyceraldehyde 3-phosphate dehydrogenase (GAPDH).
Time Frame: pre-dose, 1, 2, 4, 6, 24, and 48 hours post-dose (3 cycles)
Population: Number of participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mRNA relative values (ratio with GAPDH)
Groups:
- hENT - Cycle 1: Mean hENT expression evaluated at Cycle 1.
- hENT - Cycle 2: Mean hENT expression evaluated at Cycle 2.
- hENT - Cycle 3: Mean hENT expression evaluated at Cycle 3.
Arm/Group | hENT - Cycle 1 | hENT - Cycle 2 | hENT - Cycle 3
Number analyzed (Participants) | 19 | 19 | 19
mRNA relative values (ratio with GAPDH)
  Pre-Dose | 0.86 (0.03) | 0.86 (0.03) | 0.87 (0.02)
  1 Hour Post-Dose | 0.88 (0.04) | 0.89 (0.04) | 0.90 (0.03)
  2 Hours Post-Dose | 0.88 (0.04) | 0.90 (0.04) | 0.90 (0.04)
  4 Hours Post-Dose | 0.86 (0.04) | 0.88 (0.05) | 0.86 (0.03)
  6 Hours Post-Dose | 0.86 (0.04) | 0.86 (0.04) | 0.86 (0.02)
  24 Hours Post-Dose | 0.89 (0.04) | 0.91 (0.04) | 0.91 (0.02)
  48 Hours Post-Dose | 0.90 (0.04) | 0.91 (0.04) | 0.91 (0.02)
Statistical Analysis 1: Comparison: hENT - Cycle 1 vs hENT - Cycle 2 vs hENT - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 1 Hour Post-Dose (1 hour across cycles compared with pre-dose across cycles)
Statistical Analysis 2: Comparison: hENT - Cycle 1 vs hENT - Cycle 2 vs hENT - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 2 Hours Post-Dose (2 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 3: Comparison: hENT - Cycle 1 vs hENT - Cycle 2 vs hENT - Cycle 3; Test type: Superiority or Other; p = 0.333, Repeated Measures Analysis of Variance — P-value for 4 Hours Post-Dose (4 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 4: Comparison: hENT - Cycle 1 vs hENT - Cycle 2 vs hENT - Cycle 3; Test type: Superiority or Other; p = 0.849, Repeated Measures Analysis of Variance — P-value for 6 Hours Post-Dose (6 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 5: Comparison: hENT - Cycle 1 vs hENT - Cycle 2 vs hENT - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 24 Hours Post-Dose (24 hours across cycles compared with pre-dose across cycles)
Statistical Analysis 6: Comparison: hENT - Cycle 1 vs hENT - Cycle 2 vs hENT - Cycle 3; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis of Variance — P-value for 48 Hours Post-Dose (48 hours across cycles compared with pre-dose across cycles)

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=19)
Anaemia (Blood and lymphatic system disorders) | 5 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Arrhythmia (Cardiac disorders) | 3 (4)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7)
Asthenia (General disorders) | 9 (13)
Chest pain (General disorders) | 3 (7)
Fatigue (General disorders) | 4 (4)
General physical health deterioration (General disorders) | 3 (3)
Mucosal inflammation (General disorders) | 8 (11)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 14 (27)
Omphalitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
Transaminases (Investigations) | 2 (3)
Transaminases increased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days